CLINICAL TRIAL: NCT03877744
Title: Using Interactive Virtual Presence to Remotely Assist Parents With Child Restraint Installations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Safe Kids Worldwide (Unknown)
Responsible Party: Principal Investigator, David Schwebel, University Professor & Associate Dean, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01HD099131 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Car Seat Installation

STUDY DESIGN:
Intervention Model Description: randomized non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive virtual presence (Experimental): Participants will engage remotely with a certified child restraint technician via interactive virtual presence. They will work together to help the participant install his or her child restraint properly into his or her vehicle. Standard Safe Kids Worldwide protocols will be followed, with the exception that the interaction will occur remotely via interactive virtual presence.
  Interventions: Behavioral: interactive virtual presence
- Live technician (Active Comparator): Participants will engage live with a certified child restraint technician. They will work together to help the participant install his or her child restraint properly into his or her vehicle. Standard Safe Kids Worldwide protocols will be followed.
  Interventions: Behavioral: live technician

INTERVENTIONS:
Behavioral: interactive virtual presence — parents will install car seat through remote guidance via interactive virtual presence
  Arms: Interactive virtual presence
Behavioral: live technician — parents will install car seat through guidance from a live certified technician who is present
  Arms: Live technician

SUMMARY:
Motor vehicle crashes cause the death of an American child every 3 hours, more than any other cause. When installed correctly, car seats reduce risk of serious injury and death to infants and young children. Unfortunately, a large portion of child restraints is installed incorrectly. A network of trained technicians work across the country to assist parents in achieving correct use of child restraints through scheduled "car seat checks," where technicians work with parents to install restraints in their vehicles. Car seat checks are effective in reducing errors in child restraint installations. However, the services are highly underutilized.

The present study evaluates use of interactive virtual presence technology (also called interactive merged reality) to remotely assist parents to install child restraints correctly into their vehicles. Building from small pilot studies on the topic, the investigators will conduct a randomized non-inferiority trial to evaluate whether parents who install child restraints while communicating with a remote expert technician via interactive virtual presence achieve installations and learning that are not inferior in their safety to parents who install restraints live with a remote technician onsite.

The investigators will recruit 1476 parents at 7 locations nationwide and randomly assign consenting parents to install their child restraint either via interactive virtual presence or with a live technician. The correctness of installation safety will be assessed using objective checklists, both following installation and again four months later. The investigators aim to demonstrate that child restraint installation is accurate (>90% correct) when conducted remotely via interactive virtual presence, that such installations are not inferior to the accuracy of installation with a live on-site expert, and that parents learn and retain information about correct child restraint installation.

DETAILED DESCRIPTION:
Motor vehicle crashes cause the death of an American child every 3 hours, more than any other cause. When installed correctly, car seats (also called "child restraints") reduce risk of serious injury and death to infants and young children roughly threefold. Unfortunately, a large portion of child restraints is installed incorrectly. A network of trained technicians, many affiliated with Safe Kids Worldwide, work across the country to assist parents in achieving correct use of child restraints through scheduled "car seat checks," where technicians work with parents to install restraints in their vehicles. Car seat checks are effective in reducing errors in child restraint installations. However, the services are highly underutilized due to barriers in access, scheduling complications, and resources to staff the car seat checks sufficiently to meet demand.

The present study evaluates use of interactive virtual presence technology (also called interactive merged reality) - joint and simultaneous remote verbal and visual interaction and exposure to the same 3D stimuli - to remotely assist parents to install child restraints correctly into their vehicles. If effective, this technology could supplement or replace car seat checks, significantly reduce the number of errors made in car seat installations nationwide, and revolutionize how government, industry, and non-profit agencies help parents install restraints.

Building from small pilot studies on the topic, the investigators propose a large randomized non-inferiority trial to evaluate whether parents, including especially underserved parents in rural areas and/or of underrepresented racial or ethnic minority background, who install child restraints while communicating with a remote expert technician via interactive virtual presence achieve installations and learning that are not inferior in their safety to parents who install restraints live with a remote technician onsite. Non-inferiority trials are a type of randomized trial whereby a novel treatment (in this case, interactive virtual presence to install child restraints) is compared to an existing treatment known to be effective (in this case, live one-on-one installation of restraints) to demonstrate the novel treatment does not perform inferiorly to the existing treatment known to be effective.

To accomplish the study goals, the investigators will recruit 1476 parents at 7 Safe Kids locations nationwide and randomly assign consenting parents to install their child restraint either via interactive virtual presence or with a live technician. The correctness of installation safety will be assessed using objective checklists, both following installation and again four months later. The investigators aim to demonstrate that child restraint installation is accurate (>90% correct) when conducted remotely via interactive virtual presence, that such installations are not inferior to the accuracy of installation with a live on-site expert, and that parents learn and retain information about correct child restraint installation.

ELIGIBILITY:
Inclusion Criteria:

* own a vehicle and have a child who rides in that vehicle using a child restraint fastened with a harness.

Exclusion Criteria:

* not physically capable of installing a child restraint into a vehicle, which may exclude individuals with various disabilities.
* not able to communicate orally in English or Spanish, although significant demand for training in other languages may alter this exclusion criteria in the future

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1498 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with qualified researchers upon written request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon written request and after primary results have been accepted for publication. We will share data until they are destroyed, which is when all foreseeable use of the data has expired.
Access Criteria: Contact the PI in writing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interactive Virtual Presence | Live Technician
Started | 699 | 799
Completed | 699 | 799
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interactive Virtual Presence | Live Technician | Total
Number analyzed (Participants) | 699 | 799 | 1498
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.15 (8.13) | 34.93 (8.91) | 35.04 (8.55)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 548 | 622 | 1170
  male | 116 | 126 | 242
  non-binary | 2 | 3 | 5
  other | 1 | 2 | 3
  prefer not to answer | 3 | 1 | 4
  missing | 29 | 45 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American or Black | 85 | 113 | 198
  Asian, Asian-American, or Pacific Islander | 91 | 71 | 162
  Caucasian or White | 409 | 449 | 858
  Native American, American Indian, or Alaskan Native | 10 | 19 | 29
  Other | 38 | 53 | 91
  Prefer not to answer | 20 | 35 | 55
  Mixxing | 46 | 59 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 110 | 135 | 245
  Not Hispanic or Latino | 512 | 556 | 1068
  Prefer not to answer | 31 | 49 | 80
  Missing | 46 | 59 | 105
Region of Enrollment [Number; unit: participants]
  United States | 699 | 799 | 1498
Participants who drive a vehicle with young children [Count of Participants; unit: Participants] | 699 | 799 | 1498

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Inspection Points Correctly Installed From Pre Installation to Post Installation
Description: Percentage of inspection points in car seat installation that are correctly installed, as assessed using objective scoring scheme
Time Frame: baseline to post intervention about an hour later
Measure: Mean (Standard Deviation); unit: percentage of inspection points
Arm/Group | Interactive Virtual Presence | Live Technician
Number analyzed (Participants) | 675 | 762
percentage of inspection points | 95.78 (6.92) | 97.33 (6.12)
Statistical Analysis 1: Comparison: Interactive Virtual Presence vs Live Technician; Test type: Non-Inferiority — Non-inferiority margin of 2.5 was set prior to study initiation with a Type I error of 0.025; p = 0.0008, Mixed Models Analysis; Controls technician,site,seat type;Techn. nested in site modeled as random effect;Model allowed heterogeneous variances across arms w Kenward-Roger df; Mean Difference (Final Values) = 1.6873, 97.5% CI 1-sided [upper limit 2.1894], Standard Error of Mean 0.2558 — Mixed model allowed the arms to have unequal variance estimates. Degrees of freedom estimated using Kenward-Rogers

ADVERSE EVENTS:
Time Frame: 4 months
Description: Does not differ from clinicaltrials.gov definitions.
Arm/Group | Interactive Virtual Presence | Live Technician
All-Cause Mortality (participants affected / at risk) | 0/699 | 0/799
Serious Adverse Events (participants affected / at risk) | 0/699 | 0/799
Other Adverse Events (participants affected / at risk) | 0/699 | 0/799

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT03877744/Prot_SAP_000.pdf